CLINICAL TRIAL: NCT04267510
Title: Clinical and Molecular Aspects of Early Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0085
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Early Osteoarthritis
Keywords: genetic sequencing
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The etiology of osteoarthritis is varied, ranging from multifactorial, environmental to monogenic. In individuals in whom osteoarthritis appears earlier than in the general population, it is called early osteoarthritis. To our knowledge, there are no large-scale genetic studies on people with early osteoarthritis. The investigators therefore sought to study the causes of monogenic osteoarthritis in people suffering from early non-syndromic osteoarthritis.

Material and method From 2013 to 2019, experts in constitutional bone disease sent patients with non-syndromic early osteoarthritis for genetic analysis to our center of competence for constitutional bone diseases. The sequencing of a panel of genes was carried out by NGS.

ELIGIBILITY:
Inclusion Criteria:

- Patients with early osteoarthritis who have undergone genetic sequencing

Exclusion Criteria:

- Patients refusing to participate in research

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with early osteoarthritis who have undergone genetic sequencing
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
identification of genetic mutation | 1 day
  sequencing out by NGS
number of genetic mutation | 1 day
  sequencing out by NGS

CONTACTS AND LOCATIONS:
Overall Officials: David GENEVIEVE, Principal Investigator — Department of Medical Genetics
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC